CLINICAL TRIAL: NCT04265651
Title: Phase 2, Open-Label, Dose-Escalation and Dose-Expansion Study of Infigratinib, an FGFR 1-3-Selective Tyrosine Kinase Inhibitor, in Children With Achondroplasia: PROPEL 2
Brief Title: Study of Infigratinib in Children With Achondroplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QBGJ398-201
Record Dates: First submitted 2020-01-29; First posted 2020-02-11 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Achondroplasia
Keywords: Skeletal dysplasia; Endochondral ossification; ACH; Shortened proximal limbs; Fibroblast growth factor receptor 3; FGFR3; Endochondral bone formation; Short-limb disproportionate dwarfism; dwarfism; Bone disease; Bone diseases, developmental; Musculoskeletal diseases; Osteochondrodysplasia; Genetic diseases, inborn; Inborn
MeSH Terms: conditions — Achondroplasia; Mucopolysaccharidosis IV; Dwarfism; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Osteochondrodysplasias; Genetic Diseases, Inborn | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Infigratinib 0.016 mg/kg (Experimental): Dose Escalation:
  Infigratinib is provided as minitablets in 2 strengths: 0.1 mg and 1 mg for daily oral administration. The dose and number of minitablets/day will be calculated based on individual participant weight. Doses will be adjusted based on weight changes approximately every 3 months.
  Interventions: Drug: Infigratinib 0.016 mg/kg
- Infigratinib 0.032 mg/kg (Experimental): Dose Escalation and PK substudy:
  Infigratinib is provided as minitablets in 2 strengths: 0.1 mg and 1 mg for daily oral administration. The dose and number of minitablets/day will be calculated based on individual participant weight. Doses will be adjusted based on weight changes approximately every 3 months.
  Interventions: Drug: Infigratinib 0.032 mg/kg
- Infigratinib 0.064 mg/kg (Experimental): Dose Escalation and PK substudy:
  Infigratinib is provided as minitablets in 2 strengths: 0.1 mg and 1 mg for daily oral administration. The dose and number of minitablets/day will be calculated based on individual participant weight. Doses will be adjusted based on weight changes approximately every 3 months.
  Interventions: Drug: Infigratinib 0.064 mg/kg
- Infigratinib 0.128 mg/kg (Experimental): Dose Escalation and PK substudy:
  Infigratinib is provided as minitablets in 2 strengths: 0.1 mg and 1 mg for daily oral administration. The dose and number of minitablets/day will be calculated based on individual participant weight. Doses will be adjusted based on weight changes approximately every 3 months.
  Interventions: Drug: Infigratinib 0.128 mg/kg
- Infigratinib 0.25 mg/kg (Experimental): Dose Escalation and PK substudy:
  Infigratinib is provided as minitablets in 2 strengths: 0.1 mg and 1 mg for daily oral administration. The dose and number of minitablets/day will be calculated based on individual participant weight. Doses will be adjusted based on weight changes approximately every 3 months.
  Dose Expansion:
  Upon identification of the recommended dose from all cohorts analyzed, an expansion cohort of 20 subjects may begin enrollment to further determine safety, tolerability, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of the selected dose.
  Interventions: Drug: Infigratinib 0.25 mg/kg

INTERVENTIONS:
Drug: Infigratinib 0.016 mg/kg — Initial cohort dose of infigratinib at the protocol-specified starting dose, with subsequent cohort escalations based on protocol-specific criteria.
  Infigratinib tablets to be administered by mouth.
  Arms: Infigratinib 0.016 mg/kg
Drug: Infigratinib 0.032 mg/kg — Subsequent cohort dose escalation based on protocol-specific criteria.
  Infigratinib tablets to be administered by mouth.
  Arms: Infigratinib 0.032 mg/kg
Drug: Infigratinib 0.064 mg/kg — Subsequent cohort dose escalation based on protocol-specific criteria.
  Infigratinib tablets to be administered by mouth.
  Arms: Infigratinib 0.064 mg/kg
Drug: Infigratinib 0.128 mg/kg — Subsequent cohort dose escalation based on protocol-specific criteria.
  Infigratinib tablets to be administered by mouth.
  Arms: Infigratinib 0.128 mg/kg
Drug: Infigratinib 0.25 mg/kg — Subsequent cohort dose escalation based on protocol-specific criteria.
  Infigratinib tablets to be administered by mouth.
  Arms: Infigratinib 0.25 mg/kg

SUMMARY:
This is a Phase 2, multicenter, open-label, dose-escalation and dose-expansion study to evaluate the safety, tolerability, and efficacy of infigratinib, a fibroblast growth factor receptor (FGFR) 1-3-selective tyrosine kinase inhibitor, in children 3 to 11 years of age with Achondroplasia (ACH) who previously participated in the PROPEL study (Protocol QBGJ398-001) for at least 6 months. The study includes dose escalation with extended treatment, and dose expansion. The study also includes a PK Substudy to fully characterize the pharmacokinetics of infigratinib in children with ACH.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by participant or parent(s) or legally authorized representative (LAR) and signed informed assent by the participant (when applicable).
2. Diagnosis of ACH, documented clinically and confirmed by genetic testing.
3. At least a 6-month period of growth assessment in the PROPEL study (Protocol QBGJ398-001) before study entry.
4. Ambulatory and able to stand without assistance
5. Able to swallow oral medication.

Exclusion Criteria:

1. Hypochondroplasia or short stature condition other than ACH.
2. In females, having had their menarche.
3. Height < -2 or > +2 standard deviations for age and sex based on reference tables on growth in children with ACH.
4. Significant concurrent disease or condition that, in the view of the Investigator and/or Sponsor, would confound assessment of efficacy or safety of infigratinib.
5. Current evidence of corneal or retinal disorder/keratopathy.
6. History of malignancy.
7. Currently receiving treatment with agents that are known strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration.
8. Treatment with growth hormone, insulin-like growth factor 1 (IGF-1), or anabolic steroids in the previous 6 months or long-term treatment (>3 months) at any time.
9. Treatment with a C-type natriuretic peptide (CNP) analog, fibroblast growth factor (FGF) ligand trap, or treatment targeting FGFR inhibition at any time.
10. Regular long-term treatment (>3 weeks) with oral corticosteroids (low-dose ongoing inhaled steroid for asthma is acceptable).
11. Treatment with any other investigational product or investigational medical device for the treatment of ACH or short stature.
12. Previous limb-lengthening surgery or guided growth surgery.
13. Fracture within 12 months of screening.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) that lead to dose decrease or discontinuation | Up to 18 months
Change from baseline in annualized height velocity | Up to 18 months
PK parameters of infigratinib (Cmax- PK substudy only) | 21 days
PK parameters of infigratinib (Clast- PK substudy only) | 21 days
PK parameters of infigratinib (Tmax- PK substudy only) | 21 days
PK parameters of infigratinib (AUC24- PK substudy only) | 21 days
PK parameters of infigratinib (T1/2- PK substudy only) | 21 days
PK parameters of infigratinib (AUCinf- PK substudy only) | 21 days
PK parameters of infigratinib (CL/F- PK substudy only) | 21 days
PK parameters of infigratinib (Vz/F- PK substudy only) | 21 days
PK parameters of infigratinib (Racc- PK substudy only) | 21 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) as a measure of safety and tolerability | Up to 18 months
Absolute height velocity (annualized to cm/year), expressed numerically and as Z-score in relation to ACH and non-ACH tables | Up to 18 months
Absolute and change from baseline in weight (kg) | Up to 18 months
Absolute and change from baseline in sitting height (cm) | Up to 18 months
Absolute and change from baseline in head circumference (cm) | Up to 18 months
Absolute and change from baseline in upper and lower arm length (cm) | Up to 18 months
Absolute and change from baseline in thigh length (cm) | Up to 18 months
Absolute and change from baseline in knee height (cm) | Up to 18 months
Absolute and change from baseline in arm span (cm) | Up to 18 months
Pharmacokinetic profile of infigratinib by assessment of maximum concentration (Cmax) | Up to 18 months
Pharmacokinetic profile of infigratinib by assessment of time-to-maximum concentration (Tmax) | Up to 18 months
Changes in pharmacodynamic parameters by assessing collagen X marker | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: QED Therapeutics VP, Clinical Development, Study Director — QED Therapeutics
Locations (19):
- United States (5):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Nemours Alfred I. Dupont Hospital for Children, Wilmington, Delaware
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Murdoch Children's Hospital, Parkville, Victoria, Australia
- Stollery Children's Hospital, Edmonton, Alberta, Canada
- France (3):
  - Hopital Femme Mere Enfant, Lyon
  - Hopital Necker-Enfants Malades, Paris
  - Hopital des Enfants, Toulouse
- Spain (3):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Vithas Hospital San José, Vitoria-Gasteiz, Álava
- United Kingdom (6):
  - Sheffield Children's Hospital, Sheffield, England
  - Birmingham Children's Hospital, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Queen Elizabeth University Hospital, Glasgow
  - Evelina London Children's Hospital, London
  - Manchester University Children's Hospital, Manchester

REFERENCES:
- [Derived] Savarirayan R, De Bergua JM, Arundel P, Salles JP, Saraff V, Delgado B, Leiva-Gea A, McDevitt H, Nicolino M, Rossi M, Salcedo M, Cormier-Daire V, Skae M, Kannu P, Phillips J 3rd, Saal H, Harmatz P, Candler T, Hill D, Muslimova E, Weng R, Bai Y, Raj S, Hoover-Fong J, Irving M, Rogoff D. Oral Infigratinib Therapy in Children with Achondroplasia. N Engl J Med. 2025 Feb 27;392(9):865-874. doi: 10.1056/NEJMoa2411790. Epub 2024 Nov 18. PMID 39555818
- [Derived] Savarirayan R, De Bergua JM, Arundel P, McDevitt H, Cormier-Daire V, Saraff V, Skae M, Delgado B, Leiva-Gea A, Santos-Simarro F, Salles JP, Nicolino M, Rossi M, Kannu P, Bober MB, Phillips J 3rd, Saal H, Harmatz P, Burren C, Gotway G, Cho T, Muslimova E, Weng R, Rogoff D, Hoover-Fong J, Irving M. Infigratinib in children with achondroplasia: the PROPEL and PROPEL 2 studies. Ther Adv Musculoskelet Dis. 2022 Mar 21;14:1759720X221084848. doi: 10.1177/1759720X221084848. eCollection 2022. PMID 35342457